CLINICAL TRIAL: NCT03127371
Title: Adjunctive Nitrous Oxide to Lidocaine Anesthesia During ED Incision and Drainage of Abscess in Adults: A Randomized Controlled Trial
Brief Title: Adjunctive Nitrous Oxide During ED Incision and Drainage of Abscess
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment rate
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Emergency Medicine Foundation (Other)
Responsible Party: Principal Investigator, Joseph Herres, Research Director, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HN4861
Record Dates: First submitted 2017-03-28; First posted 2017-04-25 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Abscess
Keywords: Nitrous Oxide; Abscess; Incision and drainage
MeSH Terms: conditions — Abscess; Surgical Wound | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitrous Oxide (Experimental): Patients undergoing incision and drainage of abscess will undergo an initial medical assessment including the history, physical examination, and vital signs. The patients will then receive Nitrous Oxide gas via a gas mixer device while undergoing standard incision and drainage of cutaneous abscess using lidocaine local anesthesia administered subcutaneously. The device will mix and deliver nitrous oxide and oxygen in a 1:1 ratio, at a fixed concentration of 50%/50%. The on demand valve requires patient inspiration to trigger dosing.
  Interventions: Drug: Nitrous Oxide
- Oxygen (Experimental): Patients undergoing incision and drainage of abscess will undergo an initial medical assessment including the history, physical examination, and vital signs. The patients will then receive 100% oxygen gas via the Nitrous Oxide gas mixer device while undergoing standard incision and drainage of cutaneous abscess using lidocaine local anesthesia administered subcutaneously. The device will deliver only oxygen at a fixed concentration of 100%. The on demand valve requires patient inspiration to trigger dosing.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Nitrous Oxide — Patients undergoing incision and drainage of abscess will undergo an initial medical assessment including the history, physical examination, and vital signs. The patients will then receive Nitrous Oxide gas via a gas mixer device while undergoing standard incision and drainage of cutaneous abscess . The device will mix and deliver nitrous oxide and oxygen in a 1:1 ratio, at a fixed concentration of 50%/50%. The on demand valve requires patient inspiration to trigger dosing.
  Other Names: Sedara Gas Mixer
  Arms: Nitrous Oxide
Drug: Oxygen — Patients undergoing incision and drainage of abscess will undergo an initial medical assessment including the history, physical examination, and vital signs. The patients will then receive 100% oxygen gas via the Nitrous Oxide gas mixer device while undergoing standard incision and drainage of cutaneous abscess . The device will deliver only oxygen at a fixed concentration of 100%. The on demand valve requires patient inspiration to trigger dosing.
  Other Names: O2
  Arms: Oxygen

SUMMARY:
This study aims to describe the safety and efficacy of adjunctive nitrous oxide to lidocaine anesthesia in decreasing pain in adults during incision and drainage (I&D) of cutaneous abscesses in the emergency department (ED). Incision and drainage has been considered one of the more painful procedures performed in the ED. Standard care recommends a minimum of local anesthesia, however, there is no consensus on the appropriateness of pain management during ED painful procedures, such as incision and drainage. Oligoanalgesia continues to be a problem for ED health care providers. Despite extensive research in mechanisms of pain, factors relating to inadequate pain management, and evidence-based pain management strategies, implementation of effective pain management in the ED is still lacking. Nitrous oxide is a weak sedative agent with analgesic and anxiolytic properties. Rapid onset and short duration of action, ease of use, and favorable cardio-respiratory profile makes it an ideal agent for analgesia in the ED and may provide a novel strategy for pain management in I&D. While it has been studied an adjunct to laceration repair in children and labor in women, the use in the ED setting is not known. Adult patients capable of consenting, with simple cutaneous abscess requiring incision and drainage are the targeted population. Eligible patients who consent to the study will be randomized to one of two groups: nitrous oxide/local anesthesia or oxygen/local anesthesia. Primary endpoints assessed will be pain scores using the VAS at baseline, ten minutes after NO administration, immediately post I&D procedure, and ten minutes after procedure completion. Additionally, secondary endpoints of patient and physician procedure satisfaction scores, total time of nitrous oxide used, and presence of adverse events, including respiratory depression defined by peripheral SaO2 below 92%, ETCO2 level above 50, a rise or decrease of 10% above or below baseline, the loss of the ETCO2 waveform for more than 15 seconds. The vital signs, medical conditions, demographics, and abscess dimensions will also be collected.

DETAILED DESCRIPTION:
This study will be a prospective, randomized, double-blinded clinical trial of patients undergoing incision and drainage of abscesses in the ED of an urban, tertiary, academic medical center. Subjects will be randomized to one of two groups: 100% oxygen or 50/50 O2/Nitrous oxide while undergoing standard incision and drainage of cutaneous abscess.

Recruitment Methods

The research associates as well as the heath care team (both residents and attending physicians) will screen patients who may need incision and drainage of abscesses in the ED and may qualify for the study. Research associates will use the Cerner/AeCIS System for screening, and they will be in charge of informed consent, enrollment, placement of the capnography monitor, as well as data collection. The health care team will be in charge of the local anesthesia and incision and drainage of abscess and all other management.

Procedures Involved in the Research

Initial medical assessment will be made in accordance with established clinical procedures, including the history, physical examination, and vital signs. If by clinical assessment the patient meets eligibility criteria, then they will be approached by a research associate for enrollment in the study. After informed consent is obtained and prior to starting the procedure, standard vital sign monitoring will be placed on the patient (electrocardiogram, non-invasive blood pressure monitoring, pulse oximetry, and capnography). The Capnostream 20 ETCO2 monitor will be used as the primary device to measure ETCO2, with a nasal cannula capable of delivering supplemental oxygen and measuring ETCO2 (Oridion Medical, Needham, MA).

The SEDARA gas mixer system [Linde Gas North America LLC] will be used as our primary nitrous oxide delivery device. It will mix and deliver nitrous oxide and oxygen in a 1:1 ratio, at a fixed concentration of 50%/50%. It uses a patient driven demand valve system that is hand held. This device provides a consistent, fixed 50%/50% blend of nitrous oxide (N2O) and oxygen (O2), eliminates the need to titrate, and provides fixed concentrations for controlled and consistent dosing. The device comparator detects dosing imbalance to protect against hypoxic mixtures, it cannot deliver nitrous gas without concurrent oxygen, and the device has an anti-asphyxia valve override. The on demand valve requires patient inspiration to trigger dosing and also allows option for 100% oxygen delivery through same delivery mask. This portable device scavenges exhaled waste gases for environmental safety, as well as a key mechanism that renders the system inoperable without it for security.

After informed consent, the patient will fill out a pre procedure questionnaire and a 100 mm VAS baseline pain scale. The patient will be randomized to either the control group (100% oxygen) or treatment group (50/50) by using a randomization scheme generated using the web site Randomization.com (http://www.randomization.com). The treating physician will measure erythema and induration using a measuring tape, estimate the amount of fluctuance as small, moderate, or large, and note the location of the abscess. Once randomized, subjects will be given the mask for delivery of inhaled gas and instructed on its use, and the research associate will mark the time the patient began using the device. The SEDARA Gas Mixer will be only facing the research associate as to ensure blinding of study arm by provider and subject. The subject will be given nitrous oxide or oxygen for a minimum of 10 minutes prior to incision and drainage. The treating physician will then clean the abscess with chlorhexidine solution. The abscess will be incised with a single linear incision using a No. 11 surgical scalpel, and a cotton tipped applicator will be used to break up loculations within the abscess cavity. The method of I&D, and decision to probe to break-up loculations will be standardized, but the degree of probing, depth, and decision to pack will be left to the discretion of the treating physician. Subjects pain will be assessed using the VAS at ten minutes after NO administration but before beginning I&D, immediately post I&D procedure, and ten minutes after procedure completion.

The subject's clinical data (refer to data management) will be entered into a standardized data collection form. Study will end when the subjects recovers back to baseline. Vital signs will be flagged electronically when a physician intervenes for clinical respiratory depression. Respiratory depression will be defined as peripheral SaO2 below 92%, ETCO2 level above 50, a rise or decrease of 10% above or below baseline, the loss of the ETCO2 waveform for more than 15 seconds. Once the procedure is complete, and the patient is deemed back to their mental status baseline, they will fill out a post procedure satisfaction questionnaire. The physician will also fill out a post procedure questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or older with cutaneous abscesses located on the trunk or extremities that required I&D were approached and offered participation in the study. Need for I&D was left to discretion of treating physician.

Exclusion Criteria:

* Abscesses larger than 5 cm in any dimension
* Abscesses located on the face, neck, scalp, hands, feet, perianal, rectal, or genital areas.
* Subjects with underlying conditions that could affect ventilation, perfusion, or metabolism including intubated subjects, history of COPD, subjects with clinical signs of cardiopulmonary instability, major trauma, shock, sepsis, ASA class 3, 4, and 5.
* Those unable to provide informed consent, nursing home residents, age less than 18 years, non-English speaking, pregnant women, subjects under police custody, or physician discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in VAS pain score from baseline | Through study completion, an average of 45 minutes
  VAS measured pre-anesthesia, pre-procedure, immediately post procedure, and 10 minutes following procedure.

SECONDARY OUTCOMES:
Nitrous oxide duration | day 1
  Total number of minutes Nitrous oxide was inhaled by patients
Physician Satisfaction Survey | day 1
  Physician satisfaction with use of Nitrous oxide/Oxygen in pain control
Patient Satisfaction Survey | day 1
  Patient satisfaction with use of Nitrous oxide/Oxygen in pain control
Pulse Rate | day 1
  beats per minute
Respiratory Rate | day 1
  breaths per minute
Blood Pressure | day 1
  mmHg
Continuous Oxygen Saturation | Baseline until 10 minutes following procedure
  Oxygen saturation measured every 20 milliseconds captured by a monitoring device during study period
Continuous End tidal CO2 | Baseline until 10 minutes following procedure
  End tidal Co2 measured every 20 milliseconds captured by a monitoring device during study period

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Herres, DO, Principal Investigator — Albert Eisntein Medical Center
Locations (1):
- Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No